CLINICAL TRIAL: NCT06018922
Title: To Evaluate the Effect of a Psychological Treatment for Patients With Gaming Disorder or Hazardous Gaming.
Brief Title: Psychological Therapy for Gaming Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-06666-01; 2021-06666-01 (Other: Swedish Ethical Review Authority)
Record Dates: First submitted 2023-06-14; First posted 2023-08-31 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Gaming Disorder; Internet Gaming Disorder
Keywords: Gaming
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychological therapy for Gaming Disorder (Experimental): They will be offered a module-based psychological treatment that combines Cognitive behavioral therapy (CBT) and Family therapy (FT).
  Interventions: Behavioral: Psychological treatment

INTERVENTIONS:
Behavioral: Psychological treatment — The treatment is module-based, and the clinician are supposed to choose a small number of modules to work with depending on the patients need. The individual CBT modules are: 1) Behavioral activation, 2) Accepting thought, 3) Emotion regulation, 4) Impulse control, 5) Procrastination, 6) Relationships, 7) Problem-solving skills, 8) Structuring everyday-life, 9) Diet-Exercise-Sleep, and 10) Social anxiety. The family therapy modules are: 1) Psychoeducation about gaming, 2) Encourage other activities, 3) Positive time together, 4) Expectations and the patients abilities, 5) Making agreements in the family, 6) Emotional validation, and 7) Conflict management.

SUMMARY:
Gaming is a common leisure activity, both for children and adult, and while it is generally a positive experience for most, it can lead to problems for some individuals. There is currently a lack of knowledge of when video gaming becomes a problem and why, and there is a lack of evidence-based interventions for treating Gaming disorder. This pilot study aims to evaluate a new treatment manual for Gaming Disorder, which consists of modules based on cognitive behavioral therapy and family therapy. The therapy can be provided as individual therapy to the patient, to relatives, or as family therapy involving both the patient and their relatives. This study is an effectiveness trials and will follow all-patients at the clinic who will be offered the treatment.

The hypothesis is that the manual-based psychotherapy for Gaming Disorder will result in a reduction of Gaming Disorder symptoms and psychological distress, as well as an improvement in daily functioning.

DETAILED DESCRIPTION:
This study is a part of the clinical work at Gamingprojektet Maria Malmö, which is an outpatient clinic for patients with problematic gaming or Gaming Disorder. The clinic is focused on young people over 13 years of age and adults with problematic gaming or who meet the diagnosis of Gaming Disorder.

The study will aim to evaluate a new treatment that has been developed and are offered at Gamingprojektet Maria Malmö for patients with a problematic gaming behavior or Gaming Disorder. Before starting the treatment, they will undergo a semi-structured interview about their gaming habits, motivation for playing, demographic information, gambling, social habits, family climate, physical health, and psychiatric comorbidity. This is combined with self-assessment questionnaires on mental health, social media habits, alcohol use, drug use, gambling, emotion regulation, and everyday functioning. They will be offered a psychological treatment that combines Cognitive behavioral therapy (CBT) and Family therapy (FT). At each session, they will answer short questions about their well-being, how much they have played in the past week, and how much their well-being is related to their gaming. After completing the treatment, the patients will undergo the same semi-structured interview and questionnaires as pre-treatment. Three months after the treatment has ended, they will be called for a follow-up, where they will complete questioners about symptoms of Gaming disorder and psychological wellbeing. The study is conducted fully integrated into regular clinical practice, which allows for the feasibility and possibilities for implementation to be studied directly in connection with the study and in relation to treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Can read and speak Swedish fluidly.
* ≥ 13 years of age
* Are treatment seeking for problematic gaming or Gaming disorder

Exclusion Criteria:

- Somatic or psychiatric disease that is contraindicating or severely complicates the implementation of the intervention (e.g., ongoing psychotic, manic or hypomanic episode or neuropsychiatric condition with severe disability)

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
The Gaming Disorder Test (GDT) | At baseline (Timepoint (T) 0); Post treatment: an average of 9 months from baseline (T2); At follow up: 3 months after post treatment (T3)
  Change in symptoms of Gaming Disorder Min: 4 Max: 20 A higher outcome means worse gaming problems
Internet Gaming Disorder Scale-Short-Form (IGDS9-SF) | At baseline (Timepoint (T) 0); Post treatment: an average of 9 months from baseline (T2); At follow up: 3 months after post treatment (T3)
  Change in symptoms of Internet Gaming Disorder. Min: 9 Max: 45 A higher outcome means worse gaming problems
Time spent on gaming in the last week | At baseline (Timepoint (T) 0); Post assessment: an average of 4 weeks from baseline (T1); Post treatment: an average of 9 months from baseline (T2); At follow up: 3 months after post treatment (T3)
  Change in time spent on gaming per week
Time spent on gaming in the last week during the treatment | Once a week during the treatment period: (Post-assessment to Post-treatment) an average of 25 weeks
  Change in time spent on gaming per week during the treatment
Clinical Outcomes in Routine Evaluation - Outcome Measure 34 (Core-OM 34) | At baseline (Timepoint (T) 0); Post assessment: an average of 4 weeks from baseline (T1); Post treatment: an average of 9 months from baseline (T2); At follow up: 3 months after post treatment (T3)
  Change in self-report measure of psychological distress (for the the patients 16 years and older) Min: 0 Max: 136 A higher outcome means higher psychological distress
The Revised Child Anxiety and Depression Scale (RCADS) Youth | At baseline (Timepoint (T) 0); Post assessment: an average of 4 weeks from baseline (T1); Post treatment: an average of 9 months from baseline (T2); At follow up: 3 months after post treatment (T3)
  Change in self-report measure of psychological distress (For children) a 47-item self-report questionnaire with subscales including: separation anxiety disorder, social phobia, generalized anxiety disorder, panic disorder, obsessive compulsive disorder, and low mood.
  Min: 0 Max: 141 A higher outcome means higher psychological distress
The Revised Child Anxiety and Depression Scale (RCADS) Parent | At baseline (Timepoint (T) 0); Post assessment: an average of 4 weeks from baseline (T1); Post treatment: an average of 9 months from baseline (T2); At follow up: 3 months after post treatment (T3)
  Change in self-report measure of psychological distress (For children) a parent 47-item questionnaire about their children with subscales including: separation anxiety disorder, social phobia, generalized anxiety disorder, panic disorder, obsessive compulsive disorder, and low mood.
  Min: 0 Max: 141 A higher outcome means higher psychological distress
The Gaming Addiction Identification Test (GAIT) | At baseline (Timepoint (T) 0); Post treatment: an average of 9 months from baseline (T2); At follow up: 3 months after post treatment (T3)
  Change in a parent report measure of problematic gaming in adolescents (For children) Min: 0 Max: 35 A higher outcome means worse gaming problems

SECONDARY OUTCOMES:
Mini International Neuropsychiatric Interview (MINI) | At baseline (Timepoint (T) 0); Post treatment: an average of 9 months from baseline (T2);
  Change in if the patients meet criteria for common psychiatric diagnoses. The instrument is a brief structured diagnostic interview for the major psychiatric disorders in DSM-5. The children will be administered MINI-KID
The Global Assessment of Functioning (GAF) | At baseline (Timepoint (T) 0); Post treatment: an average of 9 months from baseline (T2);
  Change in functioning. The instrument is a numeric scale used by clinicians to rate subjectively the functioning of an patient Min: 0 Max: 100 A higher outcome means higher functioning
Working Alliance Inventory 12 (WAI) | Post treatment: an average of 9 months from baseline (T2);
  self-report questionnaire for measuring the quality of the working alliance after the treatment Min: 12 Max: 84 A higher outcome means higher working alliance
Difficulties in Emotion Regulation Scale - 16 item (Ders-16) | At baseline (Timepoint (T) 0); Post treatment: an average of 9 months from baseline (T2);
  Change in difficulties in emotion regulation Min: 16 Max: 80 A higher outcome means more problems with emotion regulation
Bergen Social Media Addiction Scale | At baseline (Timepoint (T) 0); Post treatment: an average of 9 months from baseline (T2);
  Change in symptom of social media disorder, Min: 6 Max: 30 A higher outcome means worse social media problems
Motives for Online Gaming Questionnaire (MOGQ) | At baseline (Timepoint (T) 0); Post treatment: an average of 9 months from baseline (T2);
  Change in motives for gaming. The motives are: Escape, Coping, Fantasy, Skill Development, Recreation, Competition, and Social Min: 27 Max: 135. A higher outcome indicate that the patient recognizes himself/herself to a greater extent in the various motives.
National Opinion Research Center DSM-IV Screen for Gambling: Preoccupation + Escape + Risked Relationships + Chasing (NODS-PERC) | At baseline (Timepoint (T) 0); Post treatment: an average of 9 months from baseline (T2);
  Change in symptoms of gambling disorder Min: 0 Max: 4 A higher outcome means worse gambling problems
The Alcohol Use Disorders Identification Test (Audit) | At baseline (Timepoint (T) 0); Post treatment: an average of 9 months from baseline (T2);
  Change in alcohol use Min: 0 Max: 12 A higher outcome means more problems with alcohol use
Drug Use identification list | At baseline (Timepoint (T) 0); Post treatment: an average of 9 months from baseline (T2);
  Change in drug use. By a list to identify use of common substances and frequency of use.
  Min: 0 Max: 45. A higher outcome means more problems with drug use

CONTACTS AND LOCATIONS:
Overall Officials: Emma Claesdotter-Knutsson, MD; PHD, Study Chair — Region Skåne
Locations (1):
- Region Skåne, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
After publication of data the IPD will be available at request.
Supporting Information: Study Protocol
Time Frame: After publication of data
Access Criteria: Not decided yet

REFERENCES:
- [Derived] Bore P, Nilsson S, Andersson M, Oehm K, Attvall J, Hakansson A, Claesdotter-Knutsson E. Effectiveness and Acceptability of Cognitive Behavioral Therapy and Family Therapy for Gaming Disorder: Protocol for a Nonrandomized Intervention Study of a Novel Psychological Treatment. JMIR Res Protoc. 2024 Aug 16;13:e56315. doi: 10.2196/56315. PMID 39151165